CLINICAL TRIAL: NCT05886296
Title: Evaluation of the Impact of a Pre-surgical Information Session for People Who Must Undergo Shoulder Rotator Cuff Surgery on Empowerment for Their Functional Rehabilitation Process.
Brief Title: Pre-surgical Information Session for People Who Must Undergo Shoulder Rotator Cuff Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Montserrat Grau-Pellicer, PhD, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01-23-280-028
Record Dates: First submitted 2023-05-18; First posted 2023-06-02 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Rotator Cuff Injuries; Surgery; Empowerment, Patient
MeSH Terms: conditions — Rotator Cuff Injuries; Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-surgical information session for people who must undergo shoulder rotator cuff surgery (Experimental): implementation of an information session for people who have to undergo rotator cuff surgery of the shoulder on the post-operative evolution
  Interventions: Behavioral: Evaluation of the impact of a pre-surgical information session for people who must undergo shoulder rotator cuff surgery on empowerment for their functional rehabilitation process.
- Usual care (No Intervention): Participants will undergo usual care

INTERVENTIONS:
Behavioral: Evaluation of the impact of a pre-surgical information session for people who must undergo shoulder rotator cuff surgery on empowerment for their functional rehabilitation process. — To evaluate the effect of the implementation of an information session for people who have to undergo rotator cuff surgery of the shoulder on the post-operative evolution of functionality, quality of life, empowerment and self-efficacy in the three months of the surgical intervention.
  Arms: pre-surgical information session for people who must undergo shoulder rotator cuff surgery

SUMMARY:
The shoulder is the most mobile joint in the human body. Movements are carried out in most of the activities we participate in, such as work, sports, household tasks, shopping and leisure activities. Shoulder diseases affect 21% of the western population and is one of the most frequent reasons for consultation in orthopedics and rehabilitation consultations.

Shoulder pain is in a large majority of cases related to the slope of the acromion and rotator cuff pathology, which would include the slope of the acromion syndrome. The degree of involvement can range from bursitis, tendinitis, to tendinous ruptures.

Initial treatment is usually conservative and may consist of anti-inflammatory medication and rehabilitation. When the pain is not relieved, surgery is usually recommended. Surgery for rotator cuff tears is increasingly performed minimally invasive, using arthroscopy.

Hospital admission days are currently being reduced, so many of the scheduled shoulder surgeries are performed via the Outpatient Surgery Unit. Often, users are not seen again by the surgeon until a week after the intervention. The affected person must empower themselves and participate actively and progressively in their recovery process. This process begins right after the surgical intervention. Therefore, it is very important that the person has all the necessary information about the surgical procedure that has been performed. Patient education is crucial to reduce anxiety and optimize surgical outcomes.

DETAILED DESCRIPTION:
This is a randomized clinical trial with an intervention group (IG) and a control group (CG). As participants are visited by orthopedic surgery, they are referred to rehabilitation. Once in rehabilitation and in order of arrival of the rehabilitation requests, the participants will be randomized into groups of 8 people/week in the IG and the CG. The first group of 8 people will be IG and the following week the second group of 8 people will be CG and so on until reaching the required sample.

The intervention will take place at the Rehabilitation Unit of the Consorci Sanitari de Terrassa

Participants will be anonymized and randomized into two groups: IG and CG. All participants will receive detailed information about the surgical procedure to which they will be subjected during the pre-surgical visit, carried out by the doctor specializing in orthopedic surgery. The information received will include risks and benefits and all participants will be able to ask any questions they may have. The IG will participate in an informational session prior to shoulder surgery. The session aims to: (1) Know the anatomy and functionality of the shoulder, (2) Understand why pain and functional disability appear, (3) Learn what to do to reduce symptoms, (4) Empower people to face the rehabilitation process. The CG will receive the usual rehabilitation protocol at the Consorci Sanitari de Terrassa, which begins three weeks after the surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* People who need shoulder surgery for shoulder rotator cuff pathology
* Over 18 years old
* Understand Spanish or Catalan
* Acceptance of informed consent

Exclusion Criteria:

* People who have already received previous surgery on the same shoulder
* People who have had previous infections in the same shoulder
* Neurological deficits and/or presence of tumors
* People with visual or cognitive deficits that prevent them from following the information session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Shoulder Functionality | baseline and 12 week
  Change of shoulder function from baseline to 12 weeks assessed with Constant Test (Maximum Score is 100 and it means the best function of the shoulder. Minimum Score is 0 and it means the worse function of the shoulder)

SECONDARY OUTCOMES:
Shoulder Function | baseline and 12 week
  Change of shoulder functionality from baseline to 12 weeks assessed with American Shoulder and Elbow Score (ASES Score). Maximum Score is 10 and it means the best function of the shoulder. Minimum Score is 0 and it means the worse function of the shoulder
Empowerment | baseline
  Ad-hoc self-efficacy perception questionnaire. Maximum Score is 60 and it means the best self-efficacy perception. Minimum Score is 0 and it means the worse self-efficacy perception
Participants' Quality of Life perception | baseline and 12 week
  Change of participant's Quality of life perception, assessed with the Euroquol questionnarie. Maximum Score is 25 and it means the best worse participant's Quality of Life perception. Minimum Score is 0 and it means the best participant's Quality of Life perception
Participant's satisfaction | 12 week
  Ad-hoc participant's satisfaction perception questionnaire. Maximum Score is 45 and it means the best participant's satisfaction. Minimum Score is 0 and it means the worse participant's satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fornieles-Bagur, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No